CLINICAL TRIAL: NCT07242391
Title: Menopausal Hormone Therapy And Neural Control Of Left Ventricular Function
Brief Title: Menopausal Hormone Therapy And Left Ventricular Function
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joshua M. Bock, Principal Investigator, Mayo Clinic
Other Study IDs: 25-006388
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Menopause; Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-menopausal females using menopausal hormone therapy: Post menopausal females taking a clinically prescribed menopausal hormone therapy (i.e. pill, patch, etc.)
  Interventions: Drug: Menopausal Hormone Therapy
- Post-menopausal females not using menopausal hormone therapy

INTERVENTIONS:
Drug: Menopausal Hormone Therapy — Taken in accordance with standard clinical practice, administered for a minimum duration of eight weeks.
  Groups: Post-menopausal females using menopausal hormone therapy

SUMMARY:
The purpose of this study is to compare left ventricular stroke volume and heart rate responses to bursts of SNA between PMF using, and not using, MHT.

ELIGIBILITY:
Inclusion Criteria

• >45-60< years of age

Exclusion Criteria

* Male sex
* Females between STRAW+10 stages -5 and 0
* PMF in STRAW+10 stage +2
* PMF using oral hormone therapy
* Females who entered menopause due to a surgical procedure or in response to pharmacotherapy (e.g., gonadotrophin releasing hormone agonists or chemotherapy)
* Heart disease such as hypertropic cardiomyopathy, congenital abnormalities, chronic heart failure, valve disease, and a history of myocardial infarction
* Medications that impact the central nervous system including selective serotonin reuptake inhibitors, anxiolytics, sedatives, anticholinergic agents, dopamine, amphetamines, or wake-promoting agents (e.g., modafinil). Other medications will be evaluated on an individual basis by the PI.
* Cardiovascular medications is also an exclusion criterion which includes those acting on the renin-angiotensin-aldosterone axis, adrenergic receptor antagonists, diuretics, nitrates, and calcium channel antagonists. Other medications will be evaluated on an individual basis by the PI.
* Pregnancy
* COPD
* Diabetes
* CKD
* Raynaud's phenomenon
* Sleep disorders
* Shift workers
* BMI ≥40.0kg/m2
* Use of nicotine-containing products within the two years preceding study visits
* Active cancer treatment

Ages: 45 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Study participants will be recruited from various Mayo Clinic departments/clinics located at Rochester and surrounding communities.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular stroke volume | Baseline
  Left ventricular stroke volume is the amount of blood pumped from the left ventricle per heartbeat (mL)

SECONDARY OUTCOMES:
Ventriculo-Arterial (VA) coupling | Baseline
  Ventriculo-Arterial (VA) coupling will be measured as the ratio of end-systolic elastance (Ees) to arterial elastance (Ea).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Bock, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No